CLINICAL TRIAL: NCT06917183
Title: Developing Strategies for Implementation and Use of the Operating Room Black Box (ORBB)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ganesh Sankaranarayanan, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU-2024-0975; AHRQ (Other Grant/Funding Number: 1R01HS029874-01A1)
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Demonstrate Effectiveness of Virtual Simulator in Improving OR Performance
Keywords: Virtual Reality; Simulation; OR Team Performance

STUDY DESIGN:
Intervention Model Description: An immersive virtual reality simulator designed to teach how to properly perform surgical safety checklist.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Control (No Intervention): Group 1 participants will not receive any additional training except for instutionally mandated training
- Group 2: Simulation (Experimental): Group 2 will practice on the simulator one session every day for 4 weeks.
  Interventions: Other: Training using the Immersive Multi- player Virtual Surgical Safety Checklist Training Simulator
- Group 3: Simulation with repeated reinforcement (Experimental): Group 3 participants will practice on the simulator one session every day for 4 weeks and will continue to practice on the simulator once per week for an additional two months to a total of 8 sessions.
  Interventions: Other: Training using the Immersive Multi- player Virtual Surgical Safety Checklist Training Simulator

INTERVENTIONS:
Other: Training using the Immersive Multi- player Virtual Surgical Safety Checklist Training Simulator — Training for performing surgical safety checklist for a period of 4 weeks.
  Arms: Group 2: Simulation; Group 3: Simulation with repeated reinforcement

SUMMARY:
The goal of this study is to evaluate the current use of Operating Room Black Box (ORBB)data in order to develop simulation-based training that improves intraoperative outcomes and safety, and to assess barriers and facilitators to its implementation.

There are 3 Aims for this study that the investigator will test, but the Aim that is the interventional portion of this study is only reported here in Aim 2 - Establish the validity and effectiveness of high-fidelity immersive virtual simulation-based training in improving operating room quality and safety.

DETAILED DESCRIPTION:
The study will use a mixed within and between subjects' design with two groups - control, and simulation. Due to the dedicated time needed to enroll and complete the sessions along with the need for complete novice subjects, the investigator will recruit medical students at UT Southwestern Medical Center (UTSW) from all years for the simulation group. For the Control group, the investigator will recruit participants from our OR team with a minimum of 5 years of experience at Clements University Hospital (CUH) consisting of surgeons, residents, scrub techs, circulating nurses, anesthesiologists, Certified Registered Nurse Anesthetists (CRNAs) or first assists. Subjects will be randomized into either a control group (didactic) or experimental group (didactic with virtual simulation training). Pre-test: Both groups will take a knowledge assessment test (Multiple choice) that measures baseline knowledge in performing surgical safety checklist. Immediately after that, the participants will be asked to perform the surgical safety checklist once on the simulator. For uniform standard, all participants will choose the role of a surgeon. Both groups will then complete an online introductory module on surgical safety checklists that will be speciﬁcally created for use at UTSW. Subjects in the experimental group will then practice on the simulator for 8 sessions with each session not exceeding an hour. The 8 sessions will be completed within three weeks of the pre-test. Deliberate practice will be used to achieve satisfactory scores in the training. A total of 3 scenarios, which will be selected from expert inputs and align with institute priority, will be selected for the training. Post-test: At the end of three weeks, subjects from both groups will once again take the online knowledge test followed by performing the checklists on the simulator. Transfer test: One week after post-test, subjects from both groups will perform surgical safety checklists in a simulated operating room at the UTSW Simulation Center to assess predictive validity. For other team members during the transfer test, the investigator will use the research team and volunteers from the surgical service team. The transfer test performance will be videotaped for assessment.

ELIGIBILITY:
Inclusion Criteria:

* OR service with a minimum of 5 years of experience that includes surgeons, residents, scrub techs, circulating nurses, anesthesiologists, CRNAs or first assists

Exclusion Criteria:

* OR team members (surgeons, scrub techs, circulating nurses, anesthesiologists, CRNAs or first assists) with less than 5 years of experience

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2027-02-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in surgical safety checklist performance at 1 month post intervention | Baseline, at one month post intervention
  Change in surgical safety checklist performance is assessed using the Compliance, engagement and quality scores computed automatically using the ORBB
Change in surgical safety checklist performance at 3 months post intervention | Baseline, at 3 months post intervention
  Change in surgical safety checklist performance is assessed using the Compliance, engagement and quality scores computed automatically using the ORBB
Change in surgical safety checklist performance at 5 months post intervention | Baseline, at 5 months post intervention
  Change in surgical safety checklist performance is assessed using the Compliance, engagement and quality scores computed automatically using the ORBB

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Sankaranarayanan, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No